CLINICAL TRIAL: NCT02068924
Title: Single Embryo Transfer: Comparison of Slow Freezing and Vitrification at Blastocyst Stage
Brief Title: Vitrification and Slow Freezing for Cryopreservation of Blastocyst
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0181
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: Slow freezing; Vitrification; Single embryo transfer
MeSH Terms: conditions — Infertility | interventions — Vitrification

ARMS (2):
- slow freezing (Experimental): Therefore, the aim of our study is to analyze whether extended culture of Day-2 top embryos to blastocyst-stage may improve the cumulative delivery rate in an in vitro fertilization program with Single Embryo Transfer policy in a prospective and randomized study integrating the transfer of fresh and frozen/thawed embryos using a slow freezing versus vitrification procedure.
  Interventions: Other: Slow freezing versus vitrification
- vitrification (Other): Therefore, the aim of our study is to analyze whether extended culture of Day-2 top embryos to blastocyst-stage may improve the cumulative delivery rate in an in vitro fertilization program with Single Embryo Transfer policy in a prospective and randomized study integrating the transfer of fresh and frozen/thawed embryos using a slow freezing versus vitrification procedure.
  Interventions: Other: Slow freezing versus vitrification

INTERVENTIONS:
Other: Slow freezing versus vitrification
  Other Names: Slow freezing:; G Freeze Kit Blast, Vitrolife, Suede; G-Thaw-kit Blast, Vitrolife, Suede; Vitrification:; RapidVit Blast, Vitrolife, Suede; Rapidwam Blast, Vitrolife, Suede

SUMMARY:
Improvement in the treatment of infertility by Assisted Reproductive Techniques (ART) allows single embryo transfer to be applied without compromising pregnancy rates after the first in vitro fertilization (IVF) or Intra Cytoplasmic Sperm Injection (ICSI) attempt in women less than 36 years old with good embryo quality. The policy of transferring more than one embryo after IVF or ICSI has been the main reason for the numerous twin or triple pregnancies reported in Europe and United States over the past 15 years. These multiple pregnancies are the main disadvantage of ART because of their negative impact on obstetrical, neonatal and economic outcome. In the past, embryos were replaced in the uterus on either Day-2 or 3 of development at the cleavage stage. With the development of physiologically-based sequential culture media, it has also been suggested that extending embryo culture to Day-5 in order to transfer the embryo at the blastocyst stage would enhance the likelihood of pregnancy. Nevertheless, it has been observed higher pregnancy rate after the transfer of fresh blastocyst but not after the transfer of thawed blastocyst frozen by slow freezing procedure.

However a recent embryo freezing technique (vitrification) seems to show significant higher pregnancy rates when blastocyst are frozen by this method. To our knowledge, no publications have reported the outcome of single embryo transfer at blastocyst stage by a prospective randomized and comparative study including the results of fresh and frozen/thawed blastocyst by these two methods (slow freezing vs. vitrification) in case of single embryo transfer .

Therefore, the aim of our study is to analyze whether extended culture of Day-2 top embryos to blastocyst-stage may improve the cumulative delivery rate in an in vitro fertilization program with Single Embryo Transfer policy in a prospective and randomized study integrating the transfer of fresh and frozen/thawed embryos using a slow freezing versus vitrification procedure.

DETAILED DESCRIPTION:
Improvement in the treatment of infertility by Assisted Reproductive Techniques (ART) allows single embryo transfer to be applied without compromising pregnancy rates after the first in vitro fertilization (IVF) or Intra Cytoplasmic Sperm Injection (ICSI) attempt in women less than 36 years old with good embryo quality. The policy of transferring more than one embryo after IVF or ICSI has been the main reason for the numerous twin or triple pregnancies reported in Europe and United States over the past 15 years. These multiple pregnancies are the main disadvantage of ART because of their negative impact on obstetrical, neonatal and economic outcome. In the past, embryos were replaced in the uterus on either Day-2 or 3 of development at the cleavage stage. With the development of physiologically-based sequential culture media, it has also been suggested that extending embryo culture to Day-5 in order to transfer the embryo at the blastocyst stage would enhance the likelihood of pregnancy. Nevertheless, it has been observed higher pregnancy rate after the transfer of fresh blastocyst but not after the transfer of thawed blastocyst frozen by slow freezing procedure.

However a recent embryo freezing technique (vitrification) seems to show significant higher pregnancy rates when blastocyst are frozen by this method. To our knowledge, no publications have reported the outcome of single embryo transfer at blastocyst stage by a prospective randomized and comparative study including the results of fresh and frozen/thawed blastocyst by these two methods (slow freezing vs. vitrification) in case of single embryo transfer .

Therefore, the aim of our study is to analyze whether extended culture of Day-2 top embryos to blastocyst-stage may improve the cumulative delivery rate in an in vitro fertilization program with Single Embryo Transfer policy in a prospective and randomized study integrating the transfer of fresh and frozen/thawed embryos using a slow freezing versus vitrification procedure.

ELIGIBILITY:
Inclusion Criteria:

* woman < 36 years old
* first IVF or ICSI attempt with ejaculated sperm
* at least 5 ovocytes at the pick up
* at least 3 top embryos at day-2
* at least one supernumerary blastocyst with good quality at day-5 or day-6

Exclusion Criteria:

* - woman : FSH >12UI/l
* ICSI with epididymal or testicular spermatozoa
* None supernumerary blastocyst with good quality at day-5 or day-6
* Refuse by the couple to have an embryo transfer at day-5

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative delivery rate after fresh and frozen/thawed embryo transfers | 9 months after embryo transfer

SECONDARY OUTCOMES:
Delivery rate after fresh embryo transfer | 9 months after embryo transfer
Delivery rate after transfer of frozen embryos (slow freezing) | 9 months after embryo transfer
Delivery rate after transfer of frozen embryos (vitrification) | 9 months after embryo transfer
Neonatal outcome | 9 months after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Brugnon Florence, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France